CLINICAL TRIAL: NCT07317765
Title: Research on New Methods and New Models of Rehabilitation Intervention for Cancer Patients Based on Exercise and Psychological Intervention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing HuiLongGuan Hospital (Other)
Responsible Party: Principal Investigator, Xiang Yang Zhang, Professor, Beijing HuiLongGuan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-2G-4029
Record Dates: First submitted 2025-12-09; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Other: Natural Psychotherapy
- control group (Other)
  Interventions: Other: Receive routine psychotherapy and read popular science materials related to breast cancer.

INTERVENTIONS:
Other: Natural Psychotherapy — A short-term psychological intervention of natural psychotherapy will be conducted for breast cancer patients over a five-week period, using a hybrid online and offline format. The first intervention session will be delivered offline, followed by online video-based sessions thereafter.
  Arms: intervention group
Other: Receive routine psychotherapy and read popular science materials related to breast cancer. — This intervention (routine psychotherapy plus breast cancer popular science materials) is used in control group studies for data comparison purposes, serving as a baseline to evaluate the efficacy of the experimental intervention
  Arms: control group

SUMMARY:
A Randomized Controlled Trial of Natural Psychotherapy for Intervening Negative Emotions in 100 Breast Cancer Patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed breast cancer, no distant metastasis, who have completed the perioperative period and not received subsequent treatment;
* Aged 18-59 years with an expected survival period of ≥ 1 year;
* Breast cancer patients with a self-reported depression score of ≥ 53 and/or anxiety score of ≥ 50 on self-rating scales (e.g., Self-Rating Depression Scale [SDS], Self-Rating Anxiety Scale [SAS]);
* Voluntarily participating in the study after providing informed consent and signing the informed consent form.

Exclusion Criteria:

* Patients with advanced breast cancer (stage IV with distant metastasis);
* Patients receiving other psychological interventions besides this study (e.g., individual counseling, group therapy);
* Patients with severe mental illness (e.g., schizophrenia), cognitive impairment (MMSE score < 24), heart disease, severe physical illness, other cancers, or complications;
* Patients who are unable to cooperate with psychological interventions, questionnaires, or interviews; patients who request or voluntarily withdraw from this study.

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
SAS score | 5 weeks
  Self-Rating Anxiety Scale (SAS) Score range: The total score ranges from 20 to 80 after standard conversion. Interpretation of scores: Higher scores indicate more severe anxiety symptoms; conversely, lower scores reflect milder or no anxiety symptoms.
SDS score | 5 weeks
  Self-Rating Depression Scale (SDS) Score range: The total score ranges from 20 to 80 after standard conversion. Interpretation of scores: Higher scores represent more severe depressive symptoms; on the contrary, lower scores mean less severe or no depressive symptoms.

SECONDARY OUTCOMES:
Ruminative Response Scale | 5 weeks
  Ruminative Response Scale Score Range: Total scores range from 22 to 88 Score Interpretation: Higher scores indicate more frequent and severe ruminative thinking patterns, which are associated with increased risk of negative emotional states such as depression and anxiety.
Connor-Davidson Resilience Scale | 5 weeks
  Connor-Davidson Resilience Scale Score Range: Total scores range from 0 to 100 Score Interpretation: Higher scores reflect greater psychological resilience, meaning better ability to cope with adversity, stress, and trauma.
Functional Assessment of Cancer Therapy-Breast (FACT-B) | 5 weeks
  Functional Assessment of Cancer Therapy-Breast Score Range: Total scores range from 0 to 144 Score Interpretation: Higher scores represent better health-related quality of life in breast cancer patients, covering physical well-being, social/family well-being, emotional well-being, and functional well-being specific to breast cancer.
ACC score | 5 weeks
  Acceptance and Commitment Questionnaire Score Range: Total scores range from 7 to 49 Interpretation: Higher scores indicate lower psychological flexibility

CONTACTS AND LOCATIONS:
Locations (1):
- San Huan Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Data with be available on request